CLINICAL TRIAL: NCT02836821
Title: Effect of Rifampicin on the Pharmacokinetics of Apatinib in Chinese Healthy Volunteers
Brief Title: Effect of Rifampicin on the Pharmacokinetics of Apatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-DDI-02
Record Dates: First submitted 2016-06-07; First posted 2016-07-19 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — apatinib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib (Experimental): subjects receiving a single 750 mg oral dose of apatinib mesylate tablets and wash-out for 3 days,then rifampicin capsules 600 mg/day orally for 10 days with a single 750 mg oral dose of apatinib mesylate tablets co-administered on day 8 . apatinib mesylate tablets was administered in the morning after an overnight fast of at least 10 h
  Interventions: Drug: Apatinib Mesylate Tablets; Drug: Rifampicin Capsules

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — apatinib was administered in the morning after an overnight fast of at least 10 h
  Other Names: apatinib
Drug: Rifampicin Capsules — rifampicin was administered in the morning 2 hours after breakfast
  Other Names: rifampin

SUMMARY:
The primary purpose of this study is to investigate potential pharmacokinetic interaction in healthy volunteers when apatinib is administered in combination with rifampicin. Secondary objective is evaluating the safety and tolerability of apatinib alone and when co-administered with rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* female of non-childbearing potential or male;
* age 18-45 years;
* body mass index 19-24 kg/m2 with total body weight;

Exclusion Criteria:

* clinically significant medical or surgical conditions with the potential to interfere with the absorption, distribution, metabolism or excretion of the study drugs;
* history of alcohol abuse; smoker;
* electrocardiogram(ECG) abnormality;
* blood pressure >140/90 mmHg;
* treatment with an investigational drug or any known CYP450 enzyme inducing/-inhibiting agents or herbal supplements within 14 days prior to first dose of study medication;
* Subjects were to abstain from using prescription and non-prescription drugs (other than acetaminophen as deemed necessary), vitamins and dietary supplements within 14 days prior to the first dose of study medication and throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Apatinib | 0~72h after apatinib administration

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From first administration to the seventh day after last administration
Peak Plasma Concentration (Cmax) of Apatinib | 0~72h after apatinib administration

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided